CLINICAL TRIAL: NCT04326751
Title: The Genetic Evolution and Microenvironment of Multiple Primary Lung Cancer
Brief Title: Evolution of Multiple Primary Lung Cancer (Evolution)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Guangzhou Burning Rock Medical Examination Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTHO2002
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Multiple Primary Lung Cancers; Lung Cancer; Non Small Cell Lung Cancer
Keywords: multiple primary lung cancer; ctDNA; evolution; tumor heterogeneity; microenvironment
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue and blood samples were collected from each patient. Time for blood sample collection: 1) Preoperation. 2) The 1st to 3rd day of postoperation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the evolutionary genomic landscape, explore the genetic tumor heterogeneity and microenvironment of multiple primary lung cancer (MPLC) by using tissue genetic analysis and circulating tumor DNA detection, in order to provide robust evidence for the diagnosis, treatment, and surveillance of MPLC.

DETAILED DESCRIPTION:
Multiple primary lung cancer (MPLC) has become a worldwide problem due to the difficulty in diagnosis, treatment and surveillance. Although exploring tumour clonal heterogeneity and microenvironment can help understand cancer evolution and impact therapeutic outcome, study is still lacking in this field on MPLC. Circulating tumor DNA (ctDNA) are short DNA fragments, which can be obtained conveniently and non-invasively, providing comprehensive views of the tumor as were shed by tumor cells from multiple tumor regions. Therefore, we design a prospective study of patients with surgically treated MPLC, aiming to use ctDNA technique to define the evolutionary landscape of MPLC through inter-tumor and intra-tumor heterogeneity by multi-region sampling and genetic analysis. We will also explore the the microenvironment by RNA sequencing and T cell receptor sequencing. This study may help understand the genetic evolution and microenvironment of MPLC, and provide evidence for the diagnosis, treatment and surveillance of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years

  1. Patients who are clinically diagnosed multiple lung cancers, and undergo surgical treatment.
  2. No history of any malignancy in recent 5 years.
  3. No chemotherapy, radiotherapy or targeted therapy will be performed before surgery.
  4. Surgical removal of at least 2 tumors confirmed to be lung cancer postoperatively by pathologic evaluation.

Exclusion Criteria:

1. All lesions present as pure ground-glass opacities (GGOs) on CT scans.
2. Patients who do not undergo R0 resection (including tumors located bilaterally but only unilaterally resected).
3. Unqualified blood samples.
4. Unable to comply with the study procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed multiple lung cancer patients who will receive surgical therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor heterogeneity of multiple primary lung cancer | 3 year
  Explore the intra-tumor and inter-tumor genetic heterogeneity by analysis of clonal and subclonal mutations detected by ctDNA.
Microenvironment of multiple primary lung cancer | 3 year
  Using RNA sequencing and T cell receptor (TCR) sequencing to evaluate the microenvironment of each lesion of multiple primary lung cancer, including T cell receptpr clonality ,diversity , evenness, and richness.

SECONDARY OUTCOMES:
Correlation between ctDNA and clonal variation | 3 year
  Explore the correlation between the detection rate of ctDNA and subclonal mutations of different tumor sites detected by genetic analysis.
Correlation between ctDNA and tumor burden | 3 year
  Explore the correlation between the detection rate of ctDNA and tumor burden.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.D., Study Chair — Peking University People's Hospital Thoracic Surgery Department